CLINICAL TRIAL: NCT00241592
Title: Vaporization as a Smokeless Cannabis Delivery System: A Pilot Study
Brief Title: Vaporization as a Smokeless Cannabis Delivery System
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Center for Medicinal Cannabis Research (Other)
Collaborators: University of California, San Francisco (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: C03-SF-115; CC#062; CHR# 105-22909-02; PR# 0334
Record Dates: First submitted 2005-10-18; First posted 2005-10-19 (Estimated); Last update posted 2007-06-14 (Estimated); Status verified 2007-06

CONDITIONS: Healthy Volunteers
Keywords: Cannabis; Marijuana; Vaporization; Volcano; THC
MeSH Terms: conditions — Marijuana Abuse | interventions — nabiximols

INTERVENTIONS:
Drug: Cannabis

SUMMARY:
A study to evaluate the use of a vaporization system as a smokeless delivery system for inhaled marijuana.

DETAILED DESCRIPTION:
Our primary objective is to evaluate the use of a vaporization system ( the Volcano) as a smokeless delivery system for inhaled marijuana. We will compare plasma levels of delta-9-tetrahydrocannabinol (THC), cannabinol, cannabidiol, and metabolites, including 11-OH-THC, in healthy volunteers after smoking ~400 mg each of approximately 1.8, 3.5, and 7% THC marijuana cigarettes (using the Foltin puff procedure) to those obtained when the same individuals inhale the vaporization product of the rest of the marijuana from the identical cigarette processed through the Volcano device. In addition to plasma levels, we will also compare the THC concentrations over an 8-hour time period, the subjective high experienced by the patients, and clinical evidence of cannabis effect by evaluating conjunctival hyperemia and heart rate. We will also compare the tolerability of the two methods of ingestion, and we will monitor expired carbon monoxide to evaluate whether the vaporizer reduces exposure to respiratory toxins.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-45 years Current history use of marijuana. Subjects must have smoked marijuana within the past 30 days but an amount totaling less than 10 marijuana cigarettes or the equivalent.

All men and women in this study must agree to use adequate birth control during the study. Acceptable barrier birth control methods are a male condom, female condom, diaphragm, or intra-uterine (IUD).

All women of reproductive potential (who have not reached menopause or undergone hysterectomy, oophorectomy,or tubal ligation) must have a negative urine B-HCG pregnancy test performed 48 hours before initiating the protocol-specified medication.

Able to understand and follow the instructions of the investigator and research personnel.

Able and willing to provide informed consent.

Exclusion Criteria:

* Severe coronary artery disease, uncontrolled hypertension, cardiac ventricular conduction abnormalities, or orthostatic mean blood pressure drop greater than 24mm/Hg, severe chronic obstructive pulmonary disease.

History of renal or hepatic failure. Evidence of hepatic, hematological or renal dysfunction based on judgement of physician.

Active substance abuse. Marijuana dependence as defined in DSM-IV code#304.30. Any psychiatric dysfunction that would, in the opinion of the study investigator, interfere with a participant's ability to comply with the study protocol.

Use of tobacco within the past 30 days. Subjects taking medications which may be vulnerable to drug-drug interactions such as those metabolized by the cytochrome P450 enzyme system.

Blood donation in the past 30 days. Use of smoked marijuana within 48 hours of GCRC admission. Women who are pregnant or breast-feeding may not take part in this study. Unable to read or speak English.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18
Dates: Start 2004-08; Study Completion 2005-05

PRIMARY OUTCOMES:
To assess the delivery of cannabinoids and metabolites by way of vaporization and to compare plasma levels to those obtained from smoking an identical amount of marijuana from a cigarette.

CONTACTS AND LOCATIONS:
Overall Officials: Donald I Abrams, M.D., Principal Investigator — UCSF Community Consortium
Locations (1):
- UCSF Community Consortium, San Francisco, California, United States

REFERENCES:
- [Result] Abrams DI, Vizoso HP, Shade SB, Jay C, Kelly ME, Benowitz NL. Vaporization as a smokeless cannabis delivery system: a pilot study. Clin Pharmacol Ther. 2007 Nov;82(5):572-8. doi: 10.1038/sj.clpt.6100200. Epub 2007 Apr 11. PMID 17429350
- See also: Community Consortium — http://www.communityconsortium.org
- See also: Center for Medicinal Cannabis Research — http://cmcr.ucsd.edu